CLINICAL TRIAL: NCT04108130
Title: An Anesthesia-Centered Bundle to Reduce Postoperative Pulmonary Complications: The PRIME-AIR Study
Acronym: PRIME-AIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AAAT9106; HL140177 (Other: MGH); 5UH3HL140177-03 (NIH)
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pulmonary Complications
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants in this arm will receive usual anesthetic and postoperative care as provided in each site.
- Intervention (Experimental): This arm will receive the bundle of interventions.
  Interventions: Other: Preoperative Education; Procedure: Intraoperative PEEP (Positive End-Expiratory Pressure) Individualization; Other: Individualization of Neuromuscular Blockade; Procedure: Postoperative Incentive Spirometry; Behavioral: Postoperative Ambulation

INTERVENTIONS:
Other: Preoperative Education — Brochure and video about relevance of postoperative pulmonary complications, postoperative mobilization and use of incentive spirometry.
  Arms: Intervention
Procedure: Intraoperative PEEP (Positive End-Expiratory Pressure) Individualization — PEEP will be set by maximizing respiratory system compliance along a decremental PEEP titration following an incremental recruitment maneuver.
  Arms: Intervention
Other: Individualization of Neuromuscular Blockade — Administration of neuromuscular blocking agents and their reversal will be done based on established protocol.
  Arms: Intervention
Procedure: Postoperative Incentive Spirometry — Participants will be encouraged to adhere to incentive spirometry to be started 2 hours after surgery and maintained until participant freely ambulates. Supervision will be provided 3 times/day for continuous education and management of barriers to optimal performance.
  Arms: Intervention
Behavioral: Postoperative Ambulation — Participants will be encouraged to adhere to prescription of early ambulation.
  Arms: Intervention

SUMMARY:
Postoperative pulmonary complications (PPCs) are a major cause of morbidity and mortality in surgical patients. National estimates suggest 1,062,000 PPCs per year, with 46,200 deaths, and 4.8 million additional days of hospitalization. The objective of the study is to develop and implement perioperative strategies to eliminate PPCs in abdominal surgery, the field with the largest absolute number of PPCs. We will conduct a randomized controlled pragmatic trial in 750 studied participants. The effectiveness of an individualized perioperative anesthesia-centered bundle will be compared to the usual anesthetic care in patients receiving open abdominal surgery. At the end of this project, the investigators expect to change clinical practice by establishing a new and clinically feasible anesthesia-centered strategy to reduce perioperative lung morbidity. The research will be conducted across 14 US academic centers, and will be funded by the National Institute of Health.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPCs) are a major cause of morbidity and mortality in surgical patients. National estimates suggest 1,062,000 PPCs per year, with 46,200 deaths, and 4.8 million additional days of hospitalization. Abdominal surgery is the field with the largest absolute number of PPCs. The long-term goal is to develop and implement perioperative strategies to eliminate PPCs. Whereas PPCs are as significant and lethal as cardiac complications, research in the field has received much less attention, and strategies to minimize PPCs are regrettably limited. Recently, the investigators and others have suggested a crucial role of anesthesia related interventions such as ventilatory strategies, and administration and reversal of neuromuscular blocking agents in reducing PPCs. These findings are consistent with the beneficial effects of lung protective ventilation during the adult respiratory distress syndrome (ARDS). While surgical patients differ substantially from ARDS patients as most have no or limited lung injury at the start of surgery, intraoperative anesthetic and abdominal surgery interventions result in lung derecruitment and predispose to or produce direct and indirect, potentially multiple-hit, lung injury. Thus, effective anesthetic strategies aiming at early lung protection in this group of patients are greatly needed. Indeed, the current lack of evidence results in wide and unexplained variability in anesthetic practices creating a major public health issue as some practices within usual care appear to be suboptimal and even potentially injurious. The investigators hypothesize that an anesthesia-centered bundle, based on recent findings and focused on perioperative lung protection, will minimize multiple and synergistic factors responsible for the multiple-hit perioperative pulmonary dysfunction and result in decreased incidence and severity of PPCs. Founded on strong preliminary data, we will leverage a network of US academic centers to study this hypothesis in two aims: Aim 1. To compare the number and severity of PPCs in participants receiving an individualized perioperative anesthesia-centered bundle to those in participants receiving usual anesthetic care during open abdominal surgery. For this, the investigators propose to conduct a prospective multicenter randomized controlled pragmatic trial with a blinded assessor in a total of 750 studied participants. The bundle will consist of optimal mechanical ventilation comprising individualized positive end-expiratory pressure to maximize respiratory system compliance and minimize driving pressures, individualized use of neuromuscular blocking agents and their reversal, and postoperative lung expansion and early mobilization; Aim 2. To assess the effect of the proposed bundle on plasma levels of lung injury biomarkers. The investigators theorize that our intervention will minimize overinflation and atelectasis reducing plasma levels of biomarkers of lung inflammatory, epithelial, and endothelial injury. Such mechanistic insights will facilitate bundle dissemination and support adoption as it has for lung protective ventilation for ARDS. At the end of this project, the investigators expect to change clinical practice by establishing a new and clinically feasible anesthesia-centered strategy to reduce perioperative lung morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>=18 years) scheduled for elective surgery with expected duration >=2 hours
* Open abdominal surgery including: gastric, biliary, pancreatic, hepatic, major bowel, ovarian, renal tract, bladder, prostatic, radical hysterectomy, and pelvic exenteration
* Intermediate or high risk of PPCs defined by an ARISCAT (Assess Respiratory Risk in Surgical Patients in Catalonia Score) risk score>=26

Exclusion Criteria:

* Inability or refusal to provide consent
* Inability or significant difficulty to perform any study interventions, including incentive spirometry, ambulation and/or maintaining follow-up contact with study personnel for up to 90 days after the date of surgery.
* Participation in any interventional research study within 30 days of the time of the study.
* Previous surgery within 30 days prior to this study.
* Pregnancy
* Emergency surgery
* Severe obesity (above Class I, BMI>=35 kg/m2)
* Significant lung disease: any diagnosed or treated respiratory condition that (a) requires home oxygen therapy or non-invasive ventilation (except nocturnal treatment of sleep apnea without supplemental oxygen), (b) severely limits exercise tolerance to <4 metabolic equivalents (METs) (e.g., patients unable to do light housework, walk flat at 4 miles/h or climb one flight of stairs), (c) required previous lung surgery, or (d) includes presence of severe pulmonary emphysema or bullae
* Significant heart disease: cardiac conditions that limit exercise tolerance to <4 METs
* Renal failure: peritoneal or hemodialysis requirement or preoperative creatinine >=2 mg/dL
* Neuromuscular disease that impairs ability to ventilate without assistance
* Severe chronic liver disease (Child-Turcotte-Pugh Score >9, Appendix I)
* Sepsis
* Malignancy or other irreversible condition for which 6-month mortality is estimated >=20%
* Bone marrow transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 794 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcos F Vidal Melo, MD, Principal Investigator — Columbia University
Locations (16):
- United States (16):
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - South Florida Veterans Affairs Foundation for Research and Education, Inc., Miami, Florida
  - Northwestern University, Evanston, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Hospital, Boston, Massachusetts
  - Univerisity of Massachusetts Amherst Center, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Hospital, The Bronx, New York
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
In compliance with with the NIH Policy on the Dissemination of NIH-Funded Clinical Trial Information (Notice Number NOT-OD-16-149) and NIH/NHLBI guidelines, we will submit data and specimens to the NHLBI BioLINCC (The Biologic Specimen and Data Repository Information Coordinating Center) repository, and follow procedures specified in the BioLINCC Handbook. First, list of materials to be submitted including the specimens for the NHLBI biorepository will be created. Then a data redaction plan removing personal identifiers and administrative data will be prepared, recoding low-frequency data values for subject privacy protection. The data set documentation, summary of changes made during redaction, and a summary report will be submitted to the BioLINCC repository following the standard procedures. We will comply with any modifications identified during the BioLINCC repository review, and submit the final material acceptable to the repository.
Supporting Information: Study Protocol
Time Frame: After conclusion of the study, planned for 5 years.
Access Criteria: According to the NIH/NHLBI access policies.

REFERENCES:
- [Background] PROVE Network Investigators for the Clinical Trial Network of the European Society of Anaesthesiology; Hemmes SN, Gama de Abreu M, Pelosi P, Schultz MJ. High versus low positive end-expiratory pressure during general anaesthesia for open abdominal surgery (PROVHILO trial): a multicentre randomised controlled trial. Lancet. 2014 Aug 9;384(9942):495-503. doi: 10.1016/S0140-6736(14)60416-5. Epub 2014 Jun 2. PMID 24894577
- [Background] Writing Committee for the PROBESE Collaborative Group of the PROtective VEntilation Network (PROVEnet) for the Clinical Trial Network of the European Society of Anaesthesiology; Bluth T, Serpa Neto A, Schultz MJ, Pelosi P, Gama de Abreu M; PROBESE Collaborative Group; Bluth T, Bobek I, Canet JC, Cinnella G, de Baerdemaeker L, Gama de Abreu M, Gregoretti C, Hedenstierna G, Hemmes SNT, Hiesmayr M, Hollmann MW, Jaber S, Laffey J, Licker MJ, Markstaller K, Matot I, Mills GH, Mulier JP, Pelosi P, Putensen C, Rossaint R, Schmitt J, Schultz MJ, Senturk M, Serpa Neto A, Severgnini P, Sprung J, Vidal Melo MF, Wrigge H. Effect of Intraoperative High Positive End-Expiratory Pressure (PEEP) With Recruitment Maneuvers vs Low PEEP on Postoperative Pulmonary Complications in Obese Patients: A Randomized Clinical Trial. JAMA. 2019 Jun 18;321(23):2292-2305. doi: 10.1001/jama.2019.7505. PMID 31157366
- [Background] Williams EC, Motta-Ribeiro GC, Vidal Melo MF. Driving Pressure and Transpulmonary Pressure: How Do We Guide Safe Mechanical Ventilation? Anesthesiology. 2019 Jul;131(1):155-163. doi: 10.1097/ALN.0000000000002731. PMID 31094753
- [Background] Ladha K, Vidal Melo MF, McLean DJ, Wanderer JP, Grabitz SD, Kurth T, Eikermann M. Intraoperative protective mechanical ventilation and risk of postoperative respiratory complications: hospital based registry study. BMJ. 2015 Jul 14;351:h3646. doi: 10.1136/bmj.h3646. PMID 26174419
- [Background] Wanderer JP, Ehrenfeld JM, Epstein RH, Kor DJ, Bartz RR, Fernandez-Bustamante A, Vidal Melo MF, Blum JM. Temporal trends and current practice patterns for intraoperative ventilation at U.S. academic medical centers: a retrospective study. BMC Anesthesiol. 2015 Mar 28;15:40. doi: 10.1186/s12871-015-0010-3. eCollection 2015. PMID 25852301
- [Background] de Jong MAC, Ladha KS, Vidal Melo MF, Staehr-Rye AK, Bittner EA, Kurth T, Eikermann M. Differential Effects of Intraoperative Positive End-expiratory Pressure (PEEP) on Respiratory Outcome in Major Abdominal Surgery Versus Craniotomy. Ann Surg. 2016 Aug;264(2):362-369. doi: 10.1097/SLA.0000000000001499. PMID 26496082
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] Ferrando C, Soro M, Unzueta C, Suarez-Sipmann F, Canet J, Librero J, Pozo N, Peiro S, Llombart A, Leon I, India I, Aldecoa C, Diaz-Cambronero O, Pestana D, Redondo FJ, Garutti I, Balust J, Garcia JI, Ibanez M, Granell M, Rodriguez A, Gallego L, de la Matta M, Gonzalez R, Brunelli A, Garcia J, Rovira L, Barrios F, Torres V, Hernandez S, Gracia E, Gine M, Garcia M, Garcia N, Miguel L, Sanchez S, Pineiro P, Pujol R, Garcia-Del-Valle S, Valdivia J, Hernandez MJ, Padron O, Colas A, Puig J, Azparren G, Tusman G, Villar J, Belda J; Individualized PeRioperative Open-lung VEntilation (iPROVE) Network. Individualised perioperative open-lung approach versus standard protective ventilation in abdominal surgery (iPROVE): a randomised controlled trial. Lancet Respir Med. 2018 Mar;6(3):193-203. doi: 10.1016/S2213-2600(18)30024-9. Epub 2018 Jan 19. PMID 29371130
- [Background] Brandao JC, Lessa MA, Motta-Ribeiro G, Hashimoto S, Paula LF, Torsani V, Le L, Bao X, Eikermann M, Dahl DM, Deng H, Tabatabaei S, Amato MBP, Vidal Melo MF. Global and Regional Respiratory Mechanics During Robotic-Assisted Laparoscopic Surgery: A Randomized Study. Anesth Analg. 2019 Dec;129(6):1564-1573. doi: 10.1213/ANE.0000000000004289. PMID 31743177
- [Derived] Fernandez-Bustamante A, Parker RA, Frendl G, Lee JW, Nagrebetsky A, Grecu L, Amar D, Tanaka P, Sprung J, Gupta RA, Subramanian B, Giquel J, Eikermann M, Musch G, Nadler JW, Gama de Abreu M, Bartels K, Grover M, Chen LL, Sparling J, Douin DJ, Weingarten T, Wagener G, Thompson BT, Vidal Melo MF; Perioperative Research Network (PRN) Investigators. Perioperative lung expansion and pulmonary outcomes after open abdominal surgery versus usual care in the USA (PRIME-AIR): a multicentre, randomised, controlled, phase 3 trial. Lancet Respir Med. 2025 May;13(5):447-459. doi: 10.1016/S2213-2600(25)00040-2. Epub 2025 Feb 25. PMID 40020692
- [Derived] Fernandez-Bustamante A, Parker RA, Sprung J, Eikermann M, Gama de Abreu M, Ferrando C, Thompson BT, Vidal Melo MF. An anesthesia-centered bundle to reduce postoperative pulmonary complications: The PRIME-AIR study protocol. PLoS One. 2023 Apr 6;18(4):e0283748. doi: 10.1371/journal.pone.0283748. eCollection 2023. PMID 37023031

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: This arm will receive the bundle of perioperative interventions.
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 396 | 398
Completed | 372 | 379
Not Completed | 24 | 19
Not completed — Verbal Agreement Withdrawn | 4 | 2
Not completed — Consent Withdrawn | 9 | 6
Not completed — Surgery Cancelled | 4 | 4
Not completed — Found Ineligible for Study | 4 | 3
Not completed — Consent Not Obtained for Other Reasons | 3 | 3
Not completed — Intervention Not Done and No Data Collected | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 372 | 379 | 751
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (12.0) | 61.1 (13.5) | 61.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 170 | 360
  Male | 182 | 209 | 391
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 14 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 21 | 44
  White | 278 | 294 | 572
  More than one race | 7 | 3 | 10
  Unknown or Not Reported | 43 | 47 | 90
ARISCAT Total Score [Mean (Standard Deviation); unit: score on a scale] — The Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) score is used to categorize the risk of postoperative pulmonary complications in patients undergoing non-cardiothoracic surgery. It is composed by preoperative arterial oxygen saturation, acute respiratory infection during the previous month, age, preoperative anemia, upper abdominal or intrathoracic surgery, surgical duration, and emergency surgery. Values range from a minimum of 0 to a maximum of 123, with risk categories based on the score value: low risk < 26, intermediate risk 26-44, and high risk ≥45.
  score on a scale | 40.9 (7.6) | 41.0 (7.2) | 41.0 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Postoperative Pulmonary Complications Between Participant Groups
Description: The distribution of the number and severity of accumulated post-operative pulmonary complications (PPCs) between the control and intervention groups during the first 7 days after surgery.
Time Frame: Postoperative Days 0 through 7
Population: Individual PPCs experienced by participants in both study arms.
Measure: Number; unit: complications
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
complications
  Grade 0 (none) | 84 | 73
  Grade 1 (mild) | 35 | 51
  Grade 2 (moderate) | 225 | 211
  Grade 3 (severe) | 27 | 41
  Gade 4 (ventilatory failure) | 1 | 3

2. Secondary Outcome: Number of Participants With Grade 1 and 2 Postoperative Pulmonary Complications
Description: Individual grade 3 and 4 postoperative pulmonary complications within 7 days after the day of the surgery.
Time Frame: Postoperative Days 0 through 7
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
Participants | 260 | 262

3. Secondary Outcome: Number of Participants With Grade 3 and 4 Postoperative Pulmonary Complications
Description: Individual grade 3 and 4 postoperative pulmonary complications within 7, 30, and 90 days after the day of the surgery.
Time Frame: Postoperative Days 7, 30, and 90
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
Participants
  Most Severe PPC Grade 3 or 4 by POD 7 | 28 | 44
  Most Severe PPC Grade 3 or 4 by POD 30 | 32 | 49
  Most Severe PPC Grade 3 or 4 by POD 90 | 35 | 53

4. Secondary Outcome: Number of Participants With Hypoxemia by Postoperative Day 7
Description: Presence of any hypoxemia (as defined in PPC grade 1 and 2) within 7 days after the day of the surgery.
Time Frame: Postoperative Days 0 through 7
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
Participants | 263 | 284

5. Secondary Outcome: Number of Participants With Atelectasis by Postoperative Day 7
Description: Presence of atelectasis (radiological confirmation + either temperature >37.5°C or abnormal lung symptoms/signs) by day 7 after the date of surgery.
Time Frame: Days 0 through 7 after the day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
Participants | 59 | 70

6. Secondary Outcome: Number of Participants With Pneumonia (Suspected and Proved) by Postoperative Day 7
Description: Incidence of suspected (radiological evidence without bacteriological confirmation) and proved (radiological evidence and documentation of pathological organism) pneumonia by day 7 after the date of surgery.
Time Frame: Days 0 through 7
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
Participants | 18 | 28

7. Secondary Outcome: Number of Participants With Ventilatory Dependence or Failure by Postoperative Day 7
Description: Number of participants with ventilatory dependence (Grade 3, non-invasive or invasive ventilation < 48h) or failure (Grade 4, postoperative non-invasive or invasive ventilation dependence ≥ 48h) by day 7 after the date of surgery.
Time Frame: Days 0 through 7
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
Participants | 15 | 22

8. Secondary Outcome: Length of Postoperative Oxygen Support
Description: Number of time (hours or days) spent in the postoperative oxygen therapy or other respiratory support
Time Frame: Up to 7 days post-surgery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
hours | 19.2 [4.7 to 49.4] | 14.6 [4.7 to 42.7]

9. Secondary Outcome: Number of Participants With Both Intraoperative Hypoxemia and Rescue Recruitment Maneuvers
Description: The incidence of both intraoperative hypoxemia (SpO2 < 85%) and rescue recruitment maneuvers during surgery. Received unplanned RM or PEEP titrations or adjustments during surgery for oxygenation or ventilation rescue.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
Participants | 21 | 6

10. Secondary Outcome: Number of Participants With Intraoperative Cardiovascular Events
Description: Number of participants with hypotension, bradycardia, tachycardia, arrhythmias, new ST-segment changes and cardiac arrest
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
Participants | 18 | 21

11. Secondary Outcome: Length of Hospital Stay
Description: Number of days the participant has spent in the hospital since the day of the surgery.
Time Frame: Days 0 through 7, 30, and 90
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
days | 6.8 (5.9) | 7.2 (6.1)

12. Secondary Outcome: Number of Participants With Other Hospital Readmission(s) After Initial Discharge
Description: The number of participants with hospital readmission(s), other than to the Intensive Care Unit, if admitted.
Time Frame: After the date of discharge to day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Any Major Extrapulmonary Complications
Description: Number of participants with arrhythmia, paralytic ileus, surgical site infection, infection (source uncertain), acute renal failure, and systemic inflammatory response syndrome.
Time Frame: Days 0 to 7
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 372 | 379
Participants | 43 | 48

ADVERSE EVENTS:
Time Frame: Days 0 through 7, 30, and 90. Results reported are AEs and SAEs collected by day 90.
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 5/396 | 6/398
Serious Adverse Events (participants affected / at risk) | 35/396 | 35/398
Other Adverse Events (participants affected / at risk) | 19/396 | 36/398
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=396) | Intervention (N=398)
Serious Adverse Events (General disorders) | 35 (63) | 35 (47) — Includes SAEs affecting any organ system
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=396) | Intervention (N=398)
Non-serious Adverse Events (General disorders) | 19 (44) | 36 (66) — Includes non-serious AEs affecting any organ system by day 90.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT04108130/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT04108130/SAP_001.pdf
  • Informed Consent Form (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT04108130/ICF_002.pdf